CLINICAL TRIAL: NCT05885438
Title: ACT for Healthy Living: a Brief Acceptance and Commitment Therapy Intervention for Women With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrea Davis, Graduate Student, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300010404
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will receive the ACT workshop
  Interventions: Behavioral: ACT workshop
- Waitlist Control (No Intervention): Participants in the waitlist control group will not receive the intervention until all members of the intervention group have received the workshop. Once all members of the intervention group have received the workshop, participants in the waitlist control group will be able to receive the workshop if they so desire.

INTERVENTIONS:
Behavioral: ACT workshop — This workshop is a brief behavioral intervention that teaches acceptance and commitment therapy skills (e.g., values clarification, acceptance, committed action) to approach healthy living.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to investigate if a 4-hour acceptance and commitment therapy workshop can help the adoption and maintenance of healthy lifestyle behaviors in women with obesity. The objectives are as follows:

1. To assess changes in ACT-related constructs before and after the workshop
2. To assess changes in other psychological constructs that have been shown to hinder successful weight management before and after the workshop
3. To assess changes in dietary and physical activity behaviors before and after the workshop. Participants will complete baseline questionnaires and anthropometric measures at three time points: baseline, 1 week after the workshop, and 1 month after the workshop. Researchers will compare an active intervention group to a waitlist control group to investigate the efficacy of the workshop.

DETAILED DESCRIPTION:
Acceptance and commitment therapy interventions demonstrate efficacy for weight loss. ACT-based workshops represent an innovative and potentially scalable application of this approach to obesity treatment. 70 women will be recruited to participate. Half of the participants (n = 35) will receive a brief ( approximately 4-hour) workshop that aims to facilitate the development and maintenance of healthy lifestyle behaviors using ACT principles such as valued living and committed action. Outcomes will be assessed at baseline, 1-week, and 1-month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be individuals who self-identify as women, have a BMI of >30.0 kg/m2 based on self-reported height and weight, are able to read and understand written and spoken English, and have a primary residence within 50 miles driving distance of the University of Alabama at Birmingham campus.

Exclusion Criteria:

* Exclusion criteria will include presence of eating disorder symptoms (assessed by participant self-report for a former or current diagnosis) presence of a major mood disorder (assessed by participant self-report of a current or former diagnosis), recent weight change of +/-10 pounds, recent use of prescription medication for weight loss, and current participation in another weight management program.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who self-identify as women will be eligible to participate.
Enrollment: 52 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-07-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in psychological flexibility at Week 1 | Baseline and 1 week
  The Acceptance and Action Questionnaire for Weight-Related Difficulties is a validated, self-report measure and will be used to assess change in psychological flexibility. Possible scores range from 0-22, with higher scores indicating greater psychological flexibility.
Change from baseline in distress tolerance at Week 1 | baseline and 1 week
  Distress tolerance will be measured using the Distress Tolerance Scale- Short Form (DTS), a validated, self-report measure. Possible scores range from 15 to 75, with higher scores indicating better distress tolerance
Change from baseline in valued living at Week 1 | baseline and 1 week
  The Valued Living Questionnaire is a validated, self-report measure to assess the extent to which an individual is living in a way that is consistent with their core values. Scores range from 10-100, with higher scores indicating greater consistency between values and behavior.
Change from baseline in psychological flexibility at 1 month | baseline and 1 month
  The Acceptance and Action Questionnaire for Weight-Related Difficulties is a validated, self-report measure and will be used to assess change in psychological flexibility. Possible scores range from 0-22, with higher scores indicating greater psychological flexibility.
Change from baseline in distress tolerance at 1 month | baseline and 1 month
  Distress tolerance will be measured using the Distress Tolerance Scale- Short Form (DTS), a validated, self-report measure. Possible scores range from 15 to 75, with higher scores indicating better distress tolerance
Change from baseline in valued living at 1 month | baseline and 1 month
  The Valued Living Questionnaire is a validated, self-report measure to assess the extent to which an individual is living in a way that is consistent with their core values. Scores range from 10-100, with higher scores indicating greater consistency between values and behavior.

SECONDARY OUTCOMES:
Change from baseline in weight self-stigma at Week 1 | baseline and 1 week
  Weight self-stigma will be measured using the Weight Self-Stigma Questionnaire, a validated self-report measure. This is a 23-item measure, with scores ranging from 12- 60. higher scores indicate more weight self-stigma.
Change from baseline in weight self-stigma at 1 month | baseline and 1 month
  Weight self-stigma will be measured using the Weight Self-Stigma Questionnaire, a validated self-report measure. This is a 23-item measure, with scores ranging from 12- 60. higher scores indicate more weight self-stigma.
Change from baseline in body image at Week 1 | baseline and 1 week
  Body image will be measured using the Body Shape Questionnaire, a validated, 14 item self report measure. Scores range from 14 to 84, with higher scores indicating more negative body image.
Change from baseline in body image at Month 1 | baseline and 1 month
  Body image will be measured using the Body Shape Questionnaire, a validated, 14 item self report measure. Scores range from 14 to 84, with higher scores indicating more negative body image.
Change from baseline in emotional eating at Week 1 | baseline and 1 week
  Emotional eating will be measured using the Emotional Eating Scale. This is a 25 item self-report measure with possible scores ranging from 25 to 125. Higher scores suggest greater likelihood to eat in response to emotionality.
Change from baseline in emotional eating at 1 month | baseline and 1 month
  Emotional eating will be measured using the Emotional Eating Scale. This is a 25 item self-report measure with possible scores ranging from 25 to 125. Higher scores suggest greater likelihood to eat in response to emotionality.
Change from baseline in physical activity at Week 1 | baseline and 1 week
  Physical Activity will be measured using the International Physical Activity Questionnaire -Short Form. This is a validated self report measure that provides information on frequency (times per week) and duration (minutes per session) of physical activity undertaken per week.
Change from baseline in physical activity at 1 month | baseline and 1 month
  Physical Activity will be measured using the International Physical Activity Questionnaire -Short Form. This is a validated self report measure that provides information on frequency (times per week) and duration (minutes per session) of physical activity undertaken per week.
Change from baseline in diet quality at Week 1 | baseline and 1 week
  Dietary quality will be measured using the Rapid Eating Assessment for Participants- Shortened Version (REAPS-S). The REAPS-S is a 16-item, self-report questionnaire with possible scores ranging from 16 - 48, with lower scores indicating a less healthy diet.
Change from baseline in diet quality at 1 month | baseline and 1 month
  Dietary quality will be measured using the Rapid Eating Assessment for Participants- Shortened Version (REAPS-S). The REAPS-S is a 16-item, self-report questionnaire with possible scores ranging from 16 - 48, with lower scores indicating a less healthy diet.
Change from baseline in body weight at 1 week | baseline and 1 week
  Participants will be weighed to the nearest 0.1 kg.
Change from baseline in body weight at 1 month | baseline and 1 month
  Participants will be weighed to the nearest 0.1 kg.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No